CLINICAL TRIAL: NCT05082649
Title: Investigation of Short and Long Term Results of Remote and Face-to-Face Exercise Education Programme for Chronic Low Back Pain Patients
Brief Title: Remote Exercise Programs in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aybüke Fanuscu, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-21024
Record Dates: First submitted 2021-07-14; First posted 2021-10-19 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Low Back Pain
Keywords: spinal stabilization exercise; tele-rehabilitation; low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Remotely (with video) progressive spinal stabilization exercises.
  Interventions: Other: Telerehabilitation
- Face to Face Exercises (Active Comparator): Face to face (in clinic) progressive spinal stabilization exercises.
  Interventions: Other: Face to Face Exercise

INTERVENTIONS:
Other: Face to Face Exercise — Face to face (in clinic) progressive spinal stabilization exercises.
  Arms: Face to Face Exercises
Other: Telerehabilitation — Remotely (with video) progressive spinal stabilization exercises.
  Arms: Telerehabilitation

SUMMARY:
Low back pain is a common problem that affects many people at some point in their lives. These people constitute a big part of the disease burden due to their recurrent complaints. About 45% of individuals with chronic low back pain seek medical attention. This situation makes chronic low back pain the second reason for individuals to apply to the hospital.

Exercise therapy is the first option that comes to mind in the management of low back pain. It is seen that exercise therapy both reduces the intensity of pain and reduces the recurrence rate of complaints. When the literature is examined, it is observed that among the exercise models, stabilization exercises can provide more benefits than general exercises in reducing pain and improving disability. The COVID-19 pandemic causes disruptions in face-to-face rehabilitation services. The development of telemedicine and telerehabilitation services, whose popularity is increasing with the advancing technology, gained momentum with these disruptions. With telerehabilitation, long-term treatments tailored to the needs of the patients can be offered, the cost is low, and the patients can exercise at home, on their own, at their own pace, whenever they want. These reasons make telerehabilitation stand out especially during the pandemic period. The aim of the study planned in this context is to investigate short and long-term results of remote and face-to-face exercise training on function and disease symptoms for individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Having low back pain for more than 3 months,
* Pain intensity of 3 or more according to VAS,
* literate,
* A smartphone user,
* Own a smartphone
* Individuals who are able to understand the exercises (total score >21 on the Montreal Cognitive Assessment Scale (MOCA)) will be included in the study.

Exclusion Criteria:

* Those who have been diagnosed with cervical or lumbar region pathologies,
* Cervical rapiculopathy, thoracic outlet syndrome,
* Having a malignant condition,
* Having systemic diseases such as neurological, psychological, cardiovascular, rheumatological and loss of function due to these diseases,
* History of previous surgery on the spine and upper extremity,
* Acute infection,
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-07-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of Trunk Range of Motion | 15 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline trunk range of motion at 8 weeks and 6th months
  Trunk range of motion measurement is a frequently used method in the evaluation of individuals with low back pain. Trunk range of motion measurements will be carried out before and after the exercise program using Valedo® system (Hocoma, Switzerland). Valedo® system is a professional system used in the evaluation and treatment of low back pain and valid and reliable system that is routinely used in the evaluation of trunk range of motion. Within the scope of our study, trunk flexion, extension, lateral flexion and rotation movements will be evaluated. All angles will be measured in degrees.
Evaluation of Gait Parameters - Time Characteristics 1 | 15 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline time-distance gait parameters at 8 weeks and 6th months
  Gait analyses is used to evaluate the time-distance gait parameters in chronic conditions such as low back pain. Gait analyses measurements will be carried out before and after the exercise program using OPTOGait (OPTOGait, Microgate, İtalya, 2010). The OPTOGait system consists of two bars, each 1 meter, and one a sender and the other a receiver unit. It is a portable platform that can be placed on the treadmill. Its validity and reliability have been established. During the assessment, individuals will walk in comfortable clothes and sneakers. Individuals' walking at the pace they choose will be recorded for 1 minute. Within the scope of our study, step time, gait cycle, and cadance will be evaluated and results will be recorded in seconds.
Evaluation of Gait Parameters - Time Characteristics 2 | 15 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline time-distance gait parameters at 8 weeks and 6th months
  Gait analyses is used to evaluate the time-distance gait parameters in chronic conditions such as low back pain. Gait analyses measurements will be carried out before and after the exercise program using OPTOGait (OPTOGait, Microgate, İtalya, 2010). The OPTOGait system consists of two bars, each 1 meter, and one a sender and the other a receiver unit. It is a portable platform that can be placed on the treadmill. Its validity and reliability have been established. During the assessment, individuals will walk in comfortable clothes and sneakers. Individuals' walking at the pace they choose will be recorded for 1 minute. Within the scope of our study, stance phase, swing phase, single support, double support, load response and pre-swing will be evaluated and results will be recorded as percentages.
Evaluation of Gait Parameters - Distance Characteristics | 15 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline time-distance gait parameters at 8 weeks and 6th months
  Gait analyses is used to evaluate the time-distance gait parameters in chronic conditions such as low back pain. Gait analyses measurements will be carried out before and after the exercise program using OPTOGait (OPTOGait, Microgate, İtalya, 2010). The OPTOGait system consists of two bars, each 1 meter, and one a sender and the other a receiver unit. It is a portable platform that can be placed on the treadmill. Its validity and reliability have been established. During the assessment, individuals will walk in comfortable clothes and sneakers. Individuals' walking at the pace they choose will be recorded for 1 minute. Within the scope of our study, step length and stride length will be evaluated and results will be recorded in centimeter.
Evaluation of Functional Capacity Level | 10 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline functional capacity level at 8 weeks and 6th months
  Functional capacity level will be evaluated with The Back Performance Scale. This scale is a test that evaluates the effectiveness of each activity that includes 5 different activities (socks test, gathering test, righting test, fingertip-floor test, carrying test). The Back Performance Scale test is scored between 0-15 points. A high score means poor functional capacity.
Evaluation of Pain Intensity | 5 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline pain intensity level at 8 weeks and 6th months
  Pain intensity will be evaluated with Visual Analog Scale (VAS). The VAS consists of a 10cm line. The pain experienced by the patient is marked as "0: I have no pain", "10: I have a lot of pain". Scoring is based on measuring the level marked by the participant on the line with a ruler.

SECONDARY OUTCOMES:
Evaluation of Quality of Life | 5 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline quality of life at 8 weeks and 6th months
  Quality of life will be evaluated with Nottingham Health Profile. This scale consists of 38 questions. The scale with validity and reliability has 6 subgroups: physical activity, pain, sleep, social isolation, emotional reaction and energy level. Each subgroup is scored within the range of 0-100, and a high score means poor quality of life.
Evaluation of Exercise Adaptation | 5 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline exercise adaptation at 8 weeks and 6th months
  Exercise adaptation will be evaluated with the Exercise Adherence Rating Scale (EARS). The scale consists of 3 parts. The first 2 parts of the scale consist of 6 questions and the third part consists of 10 questions. An increase in score indicates an increased adaptation to exercise. A higher score indicates greater adaptation to exercise.
Evaluation of Pain Catastrophization | 5 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline pain catastrophizing scale score at 8 weeks and 6th months
  Pain catastrophization will be evaluated with the Pain Catastrophizing Scale. Sullivan et al. was created to evaluate the catastrophic thoughts and feelings of individuals regarding the pain they feel. Consisting of 13 questions, the scale consists of rumination (thoughts spinning in the mind), magnification of pain and helplessness sub-dimensions. The total score is evaluated out of 52. A high score means a high pain catastrophe.
Evaluation of Disability | 5 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline ODI score at 8 weeks and 6th months
  Disability will be evaluated with the Oswestry Disability İndex (ODI). It was developed by Fairbank et al to evaluate the level of functional loss in individuals with low back pain. The scale consists of 10 questions about pain intensity, self-care, lifting-carrying, walking, sitting, standing, sleep, degree of change in pain, travel and social life. Each question is scored between 0-5 points. The total score is evaluated out of 100. A high score means a high level of disability.
Evaluation of Media and Social Media Usage Situations with Technological Tools | 15 minutes, through study completion, an average of 8 weeks, and 6th months after treatment, change from baseline score at 8 weeks and 6th months
  The scale was created by Rosen et al. to evaluate the use of technological tools such as computers, smart phones, and media and social media. The scale consists of two subscales and 15 factors. The factors of the usage subscale are smartphone usage, general social network usage, searching the internet, using e-mail, sharing media, using text messages (SMS), playing video games, making phone calls, watching TV, online friendship and social media friendship. The factors of the attitude subscale are positive attitude towards technology, anxiety of being without technology or technology addiction, negative attitude towards technology and transition preferences between tasks. The validity and reliability study shows that the subscales of the scale can be used together or separately. A high score means a high level of media and technology use.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)